CLINICAL TRIAL: NCT03569501
Title: Influence of DHA/Oat on Maternal and Neonatal Metabolic Health in Gestational Diabetes Mellitus
Brief Title: Impact of DHA/Oat on Metabolic Health in Gestational Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: XH-17-002
Record Dates: First submitted 2017-01-17; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-03

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: gestational diabetes mellitus; oat; docosahexaenoic acid; glycemic control; intestinal flora; newborn; leptin
MeSH Terms: conditions — Diabetes, Gestational; Gyrate Atrophy | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- nutritional guidance (No Intervention): routine care (all arms with nutritional guidance per routine care)
- oat grains (Active Comparator): 90 mg oat, per day.
  Interventions: Dietary Supplement: oat grains
- oat grains and DHA tablets (Experimental): 90 mg oat and 500 mg DHA oral tablets, per day.
  Interventions: Dietary Supplement: DHA; Dietary Supplement: oat grains
- DHA tablets (Active Comparator): 500 mg DHA oral tablets, per day.
  Interventions: Dietary Supplement: DHA

INTERVENTIONS:
Dietary Supplement: DHA — 500 mg DHA tablets
  Other Names: Docosahexaenoic acid
  Arms: DHA tablets; oat grains and DHA tablets
Dietary Supplement: oat grains — 90 mg oat, containing 4.05 mg β-glucan
  Arms: oat grains; oat grains and DHA tablets

SUMMARY:
The randomized controlled trial (RCT) recruits pregnant women with de novo diagnosis of gestational diabetes. Women bearing a singleton pregnancy are randomized into four arms: DHA, oat, oat plus DHA, and placebo. The primary outcomes are cord blood leptin concentration in the newborns and maternal fasting glucose levels at 8 weeks post-intervention.

DETAILED DESCRIPTION:
DHA is a long-chain fatty acid that has been shown to increase insulin sensitivity in basic science studies. Some studies have reported that oat (β-glucan) intake in patients with type 2 diabetes may improve glycaemic control. Evidence is emerging that gut microbiota may play an important role in energy homeostasis and glucose metabolism. This RCT aims to test the hypothesis that DHA and/or oat intake may improve glycemic control in women with gestational diabetes mellitus (GDM), and may impact metabolic health in fetuses/infants as indicated by cord blood leptin level. Changes in microbiota may be linked to these effects.

Growing evidence suggests that epigenetic changes may occur during fetal development in response to an adverse in utero environment, and this may "program" the risk of metabolic syndrome and type 2 diabetes in adulthood. GDM's offspring are programmed to be at substantially elevated risk of metabolic syndrome and type 2 diabetes in adulthood. We will explore whether the intervention may affect epigenetic profile in placental DNA in GDM.

Pregnant women bearing a singleton fetus without any evidence of malformation and with a de novo diagnosis of GDM at 22-28 weeks of gestation will be randomized into four arms: DHA, oat, oat plus DHA, and placebo. We will collect maternal blood and stool specimens on recruitment and 8-weeks post-intervention, cord blood and placenta specimens at delivery. The primary outcomes are cord blood leptin concentration in the baby, and fasting blood glucose at the 8 weeks post-intervention in the mother.

ELIGIBILITY:
Inclusion Criteria:

1. Han nationality
2. 20-45 years old
3. singleton pregnancy
4. natural conception
5. the pregnant women with de novo diagnosis of gestational diabetes mellitus during 22-28 weeks of pregnancy

Exclusion Criteria:

1. Pregnant woman or the biological father has diabetes mellitus (Type I or II)
2. the woman has severe diseases or life threatening conditions such as HIV, cancer, renal failure
3. the fetus has known congenital malformation or genetic defects
4. in-vitro fertilization
5. active hepatitis
6. tuberculosis
7. syphilis
8. drug abuser
9. multiple pregnancy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
neonatal leptin | at birth/delivery
  cord blood leptin concentration

SECONDARY OUTCOMES:
maternal fasting plasma glucose concentration | 8 weeks post-intervention
  fasting plasma glucose concentration

CONTACTS AND LOCATIONS:
Overall Officials: Yexuan Tao, Doctor, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Zhongcheng Luo, Doctor, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital Affliated to Shanghai Jiao Tong University School of Medicine;, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vandorsten JP, Dodson WC, Espeland MA, Grobman WA, Guise JM, Mercer BM, Minkoff HL, Poindexter B, Prosser LA, Sawaya GF, Scott JR, Silver RM, Smith L, Thomas A, Tita AT. NIH consensus development conference: diagnosing gestational diabetes mellitus. NIH Consens State Sci Statements. 2013 Mar 6;29(1):1-31. PMID 23748438
- [Background] Nicholson JK, Holmes E, Wilson ID. Gut microorganisms, mammalian metabolism and personalized health care. Nat Rev Microbiol. 2005 May;3(5):431-8. doi: 10.1038/nrmicro1152. PMID 15821725
- [Background] Kau AL, Ahern PP, Griffin NW, Goodman AL, Gordon JI. Human nutrition, the gut microbiome and the immune system. Nature. 2011 Jun 15;474(7351):327-36. doi: 10.1038/nature10213. PMID 21677749
- [Background] Cani PD, Geurts L, Matamoros S, Plovier H, Duparc T. Glucose metabolism: focus on gut microbiota, the endocannabinoid system and beyond. Diabetes Metab. 2014 Sep;40(4):246-57. doi: 10.1016/j.diabet.2014.02.004. Epub 2014 Mar 14. PMID 24631413
- [Background] Koren O, Goodrich JK, Cullender TC, Spor A, Laitinen K, Backhed HK, Gonzalez A, Werner JJ, Angenent LT, Knight R, Backhed F, Isolauri E, Salminen S, Ley RE. Host remodeling of the gut microbiome and metabolic changes during pregnancy. Cell. 2012 Aug 3;150(3):470-80. doi: 10.1016/j.cell.2012.07.008. PMID 22863002
- [Background] Plagemann A. Maternal diabetes and perinatal programming. Early Hum Dev. 2011 Nov;87(11):743-7. doi: 10.1016/j.earlhumdev.2011.08.018. Epub 2011 Sep 23. PMID 21945359
- [Background] Lehnen H, Zechner U, Haaf T. Epigenetics of gestational diabetes mellitus and offspring health: the time for action is in early stages of life. Mol Hum Reprod. 2013 Jul;19(7):415-22. doi: 10.1093/molehr/gat020. Epub 2013 Mar 20. PMID 23515667
- [Background] Bouchard L, Hivert MF, Guay SP, St-Pierre J, Perron P, Brisson D. Placental adiponectin gene DNA methylation levels are associated with mothers' blood glucose concentration. Diabetes. 2012 May;61(5):1272-80. doi: 10.2337/db11-1160. Epub 2012 Mar 6. PMID 22396200
- [Background] El Hajj N, Pliushch G, Schneider E, Dittrich M, Muller T, Korenkov M, Aretz M, Zechner U, Lehnen H, Haaf T. Metabolic programming of MEST DNA methylation by intrauterine exposure to gestational diabetes mellitus. Diabetes. 2013 Apr;62(4):1320-8. doi: 10.2337/db12-0289. Epub 2012 Dec 3. PMID 23209187
- [Background] Desgagne V, Hivert MF, St-Pierre J, Guay SP, Baillargeon JP, Perron P, Gaudet D, Brisson D, Bouchard L. Epigenetic dysregulation of the IGF system in placenta of newborns exposed to maternal impaired glucose tolerance. Epigenomics. 2014 Apr;6(2):193-207. doi: 10.2217/epi.14.3. PMID 24811788
- [Background] Laine R, Salminen S, Benno Y, Ouwehand AC. Performance of bifidobacteria in oat-based media. Int J Food Microbiol. 2003 May 25;83(1):105-9. doi: 10.1016/s0168-1605(02)00318-5. PMID 12672596
- [Background] Zhao JP, Levy E, Fraser WD, Julien P, Delvin E, Montoudis A, Spahis S, Garofalo C, Nuyt AM, Luo ZC. Circulating docosahexaenoic acid levels are associated with fetal insulin sensitivity. PLoS One. 2014 Jan 13;9(1):e85054. doi: 10.1371/journal.pone.0085054. eCollection 2014. PMID 24454790
- [Background] Lindsay KL, Walsh CA, Brennan L, McAuliffe FM. Probiotics in pregnancy and maternal outcomes: a systematic review. J Matern Fetal Neonatal Med. 2013 May;26(8):772-8. doi: 10.3109/14767058.2012.755166. Epub 2013 Jan 11. PMID 23205866
- [Background] Lindsay KL, Kennelly M, Culliton M, Smith T, Maguire OC, Shanahan F, Brennan L, McAuliffe FM. Probiotics in obese pregnancy do not reduce maternal fasting glucose: a double-blind, placebo-controlled, randomized trial (Probiotics in Pregnancy Study). Am J Clin Nutr. 2014 Jun;99(6):1432-9. doi: 10.3945/ajcn.113.079723. Epub 2014 Mar 19. PMID 24646819
- [Result] Shen XL, Zhao T, Zhou Y, Shi X, Zou Y, Zhao G. Effect of Oat beta-Glucan Intake on Glycaemic Control and Insulin Sensitivity of Diabetic Patients: A Meta-Analysis of Randomized Controlled Trials. Nutrients. 2016 Jan 13;8(1):39. doi: 10.3390/nu8010039. PMID 26771637
- [Result] Lindsay KL, Brennan L, Kennelly MA, Maguire OC, Smith T, Curran S, Coffey M, Foley ME, Hatunic M, Shanahan F, McAuliffe FM. Impact of probiotics in women with gestational diabetes mellitus on metabolic health: a randomized controlled trial. Am J Obstet Gynecol. 2015 Apr;212(4):496.e1-11. doi: 10.1016/j.ajog.2015.02.008. Epub 2015 Feb 14. PMID 25687568
- [Derived] Xu YJ, Wang WJ, Zhang QY, Yang MN, Zhang L, He H, Dong Y, Ouyang F, Gao Y, Zhang J, Zheng T, Luo ZC. Docosahexaenoic acid supplementation in gestational diabetes mellitus and neonatal metabolic health biomarkers. Front Nutr. 2023 Mar 20;10:1089131. doi: 10.3389/fnut.2023.1089131. eCollection 2023. PMID 37020805